CLINICAL TRIAL: NCT03693885
Title: Mild Induced Labour Prior to Planned Caesarean Delivery to Improve Neonatal and Maternal Outcome - a Randomized Trial
Brief Title: Oxytocin Administration Prior Planned Caesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: University of Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Lacarus
Record Dates: First submitted 2018-09-24; First posted 2018-10-03 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Respiratory Insufficiency Syndrome of Newborn; Breastfeeding Status
Keywords: caesarean section; Oxytocin challenge test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OCT-group (Experimental): Oxytocin challenge test: Oxytocin 5 IU/500 ml Ringer® lactate will be infused at a rate of 12 ml/h and doubled every 10 min until it induced three uterine contractions per 10-min interval at which point it will stopped.
  Interventions: Other: Oxytocin challenge test (OCT)
- Control (No Intervention): standard procedure before planned caesarean section

INTERVENTIONS:
Other: Oxytocin challenge test (OCT) — Infusion of oxytocin 5 IU/500 ml Ringer® lactate at a rate of 12 ml/h and doubled every 10 min until three uterine contractions per 10-min interval are induced, at which point it will be stopped.
  Arms: OCT-group

SUMMARY:
Spontaneous vaginal delivery of a healthy infant provokes a unique surge in stress hormone concentrations (e.g. AVP (arginine vasopressin) /copeptin) incommensurable with child or adult levels measured in any other situation. In contrast, infants delivered by primary caesarean section without preceding labour have low stress hormone concentrations at birth unless other stressors are present, including chorioamnionitis or intrauterine growth restriction. Infants delivered by caesarean section after a trial of labour show copeptin concentrations between these two extremes.

Objectives:1) To reduce neonatal respiratory morbidity and admission to the Neonatal Intensive Care Unit and increase bonding and breastfeeding by triggering uterine contractions prior to planned caesarean delivery.

2) To collect prospectively weight data of infants in the first 6 months of life to validate and expand our online neonatal weight calculator.

Study design: Open label; randomised, placebo controlled trail Intervention: Oxytocin challenge test (OCT): Infusion of oxytocin 5 IU/500 ml Ringer® lactate at a rate of 12 ml/h and doubled every 10 min until three uterine contractions per 10-min interval are induced, at which point it will be stopped.

Primary endpoint:

- Incidence of neonatal respiratory morbidity

Secondary endpoints:

* Umbilical cord blood copeptin levels
* Postnatal neonatal weight change
* Breastfeeding status

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy >34 weeks
* primary caesarean section, that is without preceding contractions or rupture of the membranes,
* absence of a contraindication to oxytocin

Exclusion Criteria:

* Chromosomal aberration
* malformation,
* IUGR,
* Nonreassuring fetal heart rate pattern,
* Placenta praevia,
* maternal substance abuse,
* infections,
* hypertension,
* preeclampsia,
* diabetes type I or II,
* autoimmune disease (antiphospholipid syndrome, lupus erythematosus, etc.),
* renal disease,
* history of more than one previous caesarean section.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1450 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of neonatal respiratory morbidity | in the first 4 hours of life
  Percentage of infants to be monitored or admitted to neonatology for respiratory distress syndrome

SECONDARY OUTCOMES:
Umbilical cord blood copeptin levels | blood sample within 30 minutes after birth
  copeptin levels in pmol/l
Postnatal neonatal weight change | postnatal day 1-4
  Maximum neonatal weight change in percent of birth weight
Breastfeeding status | 1 year
  Percentage of children who are not, partially or full breastfed

CONTACTS AND LOCATIONS:
Overall Officials: Tilo Burkhardt, MD, Principal Investigator — Dept. of Obstetrics, University Hospital Zurich
Locations (5):
- Switzerland (5):
  - University Hospital Zurich, Department of Obstetrics, Zurich, Canton of Zurich
  - Baden Cantonal Hospital, Baden
  - University Hospital Basel, Basel
  - Saint Gallen Cantonal Hospital, Sankt Gallen
  - Winterthur Cantonal Hospital, Winterthur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wellmann S, Manegold-Brauer G, Fischer T, Schaffer L, Gaertner VD, Malfertheiner SF, Burkhardt T. Improving Neonatal and Maternal Outcome by Inducing Mild Labor before Elective Cesarean Section: The Lacarus Randomized Controlled Trial. Neonatology. 2021;118(1):116-121. doi: 10.1159/000512752. Epub 2021 Jan 20. PMID 33472211